CLINICAL TRIAL: NCT06250348
Title: Exhaled Nitric Oxide : Biomarker of Acute Respiratory Distress Syndrome
Acronym: ENOBARDS
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: ENOBARDS
Record Dates: First submitted 2024-01-29; First posted 2024-02-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: ARDS, Human; Nitric Oxyde
Keywords: ARDS; Lung oedema; Capillary-alveolar permeability; Nitric Oxyde; Laser Spectroscopy
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ARDS patients: ARDS patients admitted in ICU ;intubated and mechanically ventilated for less than 24 hours
  Interventions: Other: Non invasive measure of endogenous exhaled Nitric Oxyde in exhaled gaz, by a laser spectrometer
- Control group: Healthy subjects without pulmonary nor inflammatory pathology, who underwent a benign surgical procedure (thyroid or parathyroid surgery) requiring general anesthesia with intubation and mechanical ventilation.
  Interventions: Other: Non invasive measure of endogenous exhaled Nitric Oxyde in exhaled gaz, by a laser spectrometer

INTERVENTIONS:
Other: Non invasive measure of endogenous exhaled Nitric Oxyde in exhaled gaz, by a laser spectrometer — A sample of exhaled gases is taken from the expiratory part of the respirator circuit (same way as a capnometry measurement). A laser spectrometer continuously and non-invasively monitors online the concentrations of endogenous NO exhaled by patients.

SUMMARY:
The aim of the study is to see if endogenous exhaled Nitric Oxyde (eNO) concentrations measured are significantly higher in ARDS patients admitted in ICU ; compared to control subjects in good health with no lung disease or global inflammation, operated under general anesthesia (i.e. intubated and ventilated) for thyroid or parathyroid.

DETAILED DESCRIPTION:
The measurement of endogenous exhaled NO is monitored using a laser spectrometer machine connected to the expiratory circuit of the respirator. The measure is non-invasive and made by sampling expiratory gaz like for capnography.

In control subjects, the measurement period corresponds to the first ten minutes after induction of anesthesia (with intubation) before surgical incision.

In ARDS patients in intensive care, the measurement of eNO is made in the first twenty-four hours after intubation and ventilation of the patient with mechanical respirator.

The primary endpoint is a significantly higher eNO concentration in patients suffering from Acute Respiratory Distress Syndrome (ARDS).

Secondary endpoints will assess correlations between eNO concentrations and usual ARDS severity criteria: PaO2/FiO2; ventilator-free days; length of stay in intensive care and all-cause hospital mortality at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* For ARDS patients :

  * Patients with ARDS (according to the Berlin criteria) admitted in intensive care unit and intubated for less than 24 hours.
* For control patients :

  * Patients with no major disease (classified 1 or 2 in the classification of the American Society of Anaesthesiology)
  * Patients undergoing general anaesthesia for a thyroïd or parathyroïd surgery

Exclusion Criteria:

* Minors under the age of 18 years old
* Pregnant women
* prisoners
* patients who have withdrawn their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients (from any cause) in ICU Control group : healthy patients (ASA I or II) operated for a minor surgery (thyroid or parathyroid)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Endogenous exhaled Nitric Oxyde (eNO) | Measurement of eNO over a period of 10 minutes just after induction of anesthesia
  The primary endpoint is a significantly higher eNO concentration in ARDS patients.

SECONDARY OUTCOMES:
Secondary endpoints will assess correlations between eNO concentrations and usual ARDS severity criteria | Measurement of eNO over a period of 10 minutes within the first 24 hours after intubation
  ARDS severity criteria are: Partial arterial pressure of oxygen divided by inspired fraction of oxygen (PaO2/FiO2); ventilator-free days; length of stay in intensive care and all-cause hospital mortality at 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael BRIOT, MD ; PhD, Principal Investigator — Laboratoire TIMC - Team PRETA UMR CNRS-UGA 5525 ; Grenoble Alpes University
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No
In this single-center observational study, anonymized data are collected and centralized by the principal investigator before being analyzed by the team of statisticians.

REFERENCES:
- [Background] Chollier T, Richard L, Romanini D, Brouta A, Martin JL, Moro C, Briot R, Ventrillard I. Monitoring of endogenous nitric oxide exhaled by pig lungs during ex-vivo lung perfusion. J Breath Res. 2021 Feb 11;15(2). doi: 10.1088/1752-7163/abde95. PMID 33477122